CLINICAL TRIAL: NCT03479684
Title: Randomized Trial of Genotype-guided Versus Standard for Warfarin Dosing
Brief Title: Genotype-guided Versus Standard for Warfarin Dosing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Lu Hua, chief physician of Thrombosis and Vascular Medicine Center Fuwai Hospitai, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z171100001017216
Record Dates: First submitted 2018-02-27; First posted 2018-03-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Atrial Fibrillation; Valvular Heart Disease
Keywords: warfarin; gene
MeSH Terms: conditions — Atrial Fibrillation; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gene-directed group (Experimental): the first day given model prediction dose * 1.5 times（<6mg）；the second day given model prediction dose；adjusted dose based on INR from the third day
  Interventions: Other: Gene-directed dosage of warfarin
- Standard care group (Active Comparator): the first day given 4.5mg; adjusted dose based on INR from the second day
  Interventions: Other: standard dosage of warfarin

INTERVENTIONS:
Other: Gene-directed dosage of warfarin — the first day given model prediction dose * 1.5 times（<6mg）；the second day given model prediction dose；adjusted dose based on INR from the third day
  Arms: Gene-directed group
Other: standard dosage of warfarin — the first day given 4.5mg; adjusted dose based on INR from the second day
  Arms: Standard care group

SUMMARY:
To compare the efficiency and safety between gene-oriented group and standard care group during 90 days of initial warfarin-treatment for requiring anticoagulation patients with valve replacement or atrial fibrillation with or without valvular heart disease。

DETAILED DESCRIPTION:
Due to narrow therapeutic window, and individual differences in dosage, inappropriate use of warfarin may lead to serious complications and ineffective. Based on the results of the research on the transformation of warfarin pharmacogenomics, this study investigates the clinical application of gene-directed warfarin dose prediction model through the preset dosage regimen of warfarin during the initial treatment phase. Compared with the conventional treatment, that is to say empirical medication, this study is to verify the feasibility and value of gene-oriented warfarin dose prediction model, in order to establish a practical guidance to optimize the rational use of warfarin treatment program, to enable patients to obtain effective, safe warfarin dose, and to achieve the established anticoagulant strength faster and safer, as the same time, to reduce the times of patients was blood and the incidence of bleeding/embolism, and to save costs and ensure the safety of warfarin clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years old, requiring anticoagulation because of valvular or non-valvular atrial fibrillation or after valvular replacement. Patients could visit to be followed up in our hospital clinic regularly and agree to participate in the clinical trial and sign a written informed consent.

Exclusion Criteria:

* Patients will be excluded from the trial if aged <18 years old or > 75 years old, pregnant and lactating, if treated tricuspid valve replacement, or coronary artery bypass grafting before, if diagnosed with congenital heart disease, if known their CYP2C9 or VKORC1 genotype, if taken dicoumarol drugs previously or taking them now, if not suitable for enrollment judged by researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
therapeutic INR range (TTR) 90 | at Day90
  The percentage of time in therapeutic INR range (TTR) using the number of INRs within the therapeutic range divided by the number of INRs collected, will be assessed at Day90, and the TTR of all patients will be reported.

SECONDARY OUTCOMES:
therapeutic INR range (TTR) 28 | at Day28
  The percentage of time in therapeutic INR range (TTR) using the number of INRs within the therapeutic range divided by the number of INRs collected, will be assessed at Day28, and the TTR of all patients will be reported.
Time of the first time of the target INR | 90 days
  Time of the first time for participants to reach the target INR will be collected and reported during the study.

OTHER OUTCOMES:
thrombus or embolism or bleeding complications | 90 days
  The number of thrombus or embolism or any hemorrhage events for participants through the study completion will be collected and assessed at Day90.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, MD. PhD, Principal Investigator — Thrombosis and Vascular Medicine Center
Locations (1):
- Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Consent for sharing of non identifiable study data for regulatory authorities.